CLINICAL TRIAL: NCT02534220
Title: Gingival Margin Stability After Mucogingival Plastic Surgery. The Effect of Manual Versus Powered Toothbrushing: a Randomized Clinical Trial
Brief Title: Manual Versus Oscillating-rotating Toothbrushes After Root Coverage Procedure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Milan (Other)
Responsible Party: Principal Investigator, Giulio Rasperini, Prof., University of Milan
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Oral-B
Record Dates: First submitted 2015-08-21; First posted 2015-08-27 (Estimated); Last update posted 2015-08-27 (Estimated); Status verified 2015-08

CONDITIONS: Gingival Recession
Keywords: Toothbrushing; Oral hygiene; Dental hygiene
MeSH Terms: conditions — Gingival Recession

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Manual Toothbrush (Active Comparator): Patients were instructed in the Roll Brushing Technique, twice daily for 2 min.
  Interventions: Device: Manual Toothbrush
- Oscillating-rotating toothbrush (Experimental): Patients received manufacturer's instructions for use, including brushing twice daily for 2 min.
  Interventions: Device: Oscillating-rotating toothbrush

INTERVENTIONS:
Device: Manual Toothbrush — Gum Delicate Post-Surgical Toothbrush, Oral-B, Procter & Gamble, Cincinnati, OH
  Arms: Manual Toothbrush
Device: Oscillating-rotating toothbrush — Triumph 5000, Oral-B, Procter & Gamble, Cincinnati, OH
  Arms: Oscillating-rotating toothbrush

SUMMARY:
The aim of this study is to evaluate the gingival margin stability with the use of oscillating-rotating toothbrushes compared to manual toothbrushes.

DETAILED DESCRIPTION:
BACKGROUND Oscillating-rotating power toothbrushes have been proven clinically efficacious. To the investigators' knowledge, a clinical evaluation of the safety of these toothbrushes after surgical root coverage procedure have not been published. The aim of this study is to evaluate the gingival margin stability with the use of oscillating-rotating toothbrushes compared to manual toothbrushes.

METHODS Sixty healthy patients with at least a single Miller Class I or II gingival recession underwent surgical root coverage procedure. Soft-bristle manual and powered toothbrushes were given to participants randomly assigned to control and test group, respectively. Full-mouth plaque score, Full-mouth Bleeding Score, Probing Pocket Depth and Recession Depth were recorded 1, 3 and 6 months after completion of surgical procedure. Longitudinal analyses were performed using linear random-intercept models to take into account within-subject correlations over time. Temporal trend differences across treatments by including treatment-time interaction terms were then tested using a global Wald test.

ELIGIBILITY:
Inclusion Criteria:

* Full-Mouth Plaque Score (FMPS) ≤25%
* Full-Mouth Bleeding Score (FMBS) ≤25%
* Miller Class I and II buccal recession ≥2 mm

Exclusion Criteria:

* Relevant systemic condition or disease
* Smokers
* Teeth with prosthetic crowns or restorations in the cervical area
* Presence of pulling frenum in the keratinized tissue
* Previous mucogingival or periodontal surgery in the experimental site

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2014-02; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Change in Complete Root Coverage Rate | Change in Complete Root Coverage Rate at 1 month
  Abscence of exposed root surface measured ad percentage
Change in Complete Root Coverage Rate | Change in Complete Root Coverage Rate at 3 months
  Abscence of exposed root surface measured ad percentage
Change in Complete Root Coverage Rate | Change in Complete Root Coverage Rate at 6 months
  Abscence of exposed root surface measured ad percentage

SECONDARY OUTCOMES:
Change in Recession Depth | Baseline, 1 month, 3 months, 6 months
  Distance from the gingival margin to the cementum-enamel junction, measured in millimeters
Change in Clinical Attachment Level | Baseline, 1 month, 3 months, 6 months
  Distance from the cementum-enamel junction to the bottom of the periodontal Pocket, measured in millimeters
Change in Probing Pocket Depth | Baseline, 1 month, 3 months, 6 months
  Distance from the gingival margin to the bottom of the periodontal pocket, measured in millimeters

CONTACTS AND LOCATIONS:
Overall Officials: Giulio Rasperini, Study Director — Unit of Periodontology, Department of Biomedical, Surgical and Dental Sciences, University of Milan, Foundation IRCCS Ca' Granda Policlinic
Locations (1):
- Clinica Odontoiatrica IRCCS Ospedale Maggiore Policlinico, Milan, MI, Italy